CLINICAL TRIAL: NCT03887169
Title: Oral or Enteral Administration of Methionine in Patients With Pulmonary Alveolar Proteinosis by Mutation of the MARS Gene.
Brief Title: Administration of Methionine in Patients With Pulmonary Alveolar Proteinosis by Mutation of the MARS Gene.
Acronym: MetPAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC20180338; 2018-004140-28 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Alveolar Proteinosis; Mutation Ala393Thr of the MARS Gene; mutationSer567Leu of the MARS Gene
Keywords: Pulmonary alveolar proteinosis; MARS gene; methionine
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis | interventions — Methionine; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methionine (Experimental)
  Interventions: Drug: Methionine; Drug: Vitamin B12, B9, B6, C supplementation; Diagnostic Test: Methionine/homocysteine Dosage; Diagnostic Test: Thoracic CT scan; Diagnostic Test: Abdominal and liver ultrasound.; Diagnostic Test: Brain MRI

INTERVENTIONS:
Drug: Methionine — Administration of methionine from D1 to D60
Drug: Vitamin B12, B9, B6, C supplementation — In case of hyperhomocysteinemia
Diagnostic Test: Methionine/homocysteine Dosage — Plasma concentration control of methionine and homocysteine from D0 to D75
Diagnostic Test: Thoracic CT scan — At D60
Diagnostic Test: Abdominal and liver ultrasound. — At D60
Diagnostic Test: Brain MRI — In case of abnormal neurological examination

SUMMARY:
The purpose of this study is to determine the safety and tolerance of an oral administration of methionine in the treatment of pulmonary alveolar proteinosis due to the double mutation Ala393Thr / Ser567Leu in the MARS gene. This disease is very severe and especially leads to chronic respiratory insufficiency. There is no curative treatment for this disease. The MARS gene encodes the methionine tRNA synthetase (MetRS). Mutations in this gene leads to a defect in MetRS function. In cultured mutated yeast, addition of methionine in culture medium restores MetRS function. Therefore, the investigators hypothesized that treatment of patients with methionine could have beneficial effects on the disease.

DETAILED DESCRIPTION:
Pulmonary alveolar proteinosis (PAP) is a rare respiratory disorder. Recently, a genetic cause has been identified for a specific form of PAP predominant on La Reunion Island. This form is characterized by a multisystem phenotype including PAP, failure to thrive, hepatic involvement and chronic inflammation. This is a severe disease without any specific treatment and a high rate of mortality related to end-stage respiratory insufficiency. Two recurrent mutations were isolated in the MARS gene that encodes the methionine tRNA synthetase (MetRS). This enzyme catalyzes the ligation of methionine to tRNA and is critical for protein biosynthesis. Functional studies on mutated yeast show an altered growth and protein synthesis as compared to control yeast. Addition of methionine in culture medium corrects these defects. Complementary experiments on human purified MetRS show altered enzymatic catalytic parameters in mutated forms. Increasing blood concentration of methionine in patients could correct these parameters and potentially improve patients' phenotype in this severe disorder where no curative treatment exists.

The main objective of this protocol is to determine the tolerance of a prolonged daily supplementation of methionine in patients presenting a MARS related PAP. The secondary objectives are to determine the efficiency of such treatment on respiratory, hepatic, inflammatory and growth status.

To meet the objectives of the study, enrolled patients will receive daily oral or enteral methionine administration at increasing doses, under surveillance of plasma levels of methionine and homocysteine, and possible clinical side effects, until determining the "ideal" dose for each patient.

Once daily dosage determined for each patient, this dosage will be continued for a total of 2 months with daily clinical monitoring of tolerance and bi-monthly plasma levels surveillance of methionine and homocysteine.

ELIGIBILITY:
Inclusion Criteria:

* Minor Patient with alveolar proteinosis by double mutation Ala393Thr and SER567LEU of the MARS gene, genetically proven.
* Patient in need of prolonged hospitalization in Necker for treatment of bronchial-alveolar washes in the context of care.
* Patient for which methionine can be administered orally or by enteral probe (Nasogastric or gastrostomy probe)
* Signed Informed consent form by parents / legal guardian

Exclusion Criteria:

* Patient with alveolar proteinosis by other mutations of the MARS gene
* Patient with alveolar proteinosis secondary to another etiology or without identified cause
* Refusal to participate in the study
* High blood pressure requiring drug treatment
* Heart failure
* Known hypersensitivity to one of the substances used or potentially used in the study: methionine, vitamins B6, B12, B9 and C
* Pre-Hypermethioninemia (Methioninemia > + 2 DS of normal for age) whatever the cause

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Tolerance Assessment | From day 0 to day 75
  No adverse event from day 0 to day 75.

SECONDARY OUTCOMES:
Respiratory rate (cycles /min) | At day 0, day 15, day 30, day 45, day 60, day 75
  number of cycles per minute
Oxygen need (L/min) | At day 0, day 15, day 30, day 45, day 60, day 75
  Flow in L/min
Respiratory signs of struggle | At day 0, day 15, day 30, day 45, day 60, day 75
  Presence or absence of signs
Lung lesions | At Day 60
  Lesions appearance on thoracic CT scan, scored form 0 to 4
Lipo-proteinaceous material | At each bronchial-alveolar washes during the 2,5 months
  Fluid examination
Weight | At Day 15, Day 30, Day 45, Day 60, Day 75
  To evaluate Nutritional status
mid upper arm circumference / head circumference rapport | At Day 15, Day 30, Day 45, Day 60, Day 75
  To evaluate Nutritional status
Hepatomegaly | At Day 0, Day 15, Day 30, Day 45, Day 60, Day 75
  liver damage evaluate by physician during clinical examination
cholestasis and hepatic cytolysis | At Day 0, Day 15, Day 30, Day 60, Day 75
  liver damage evaluate by biological parameters : ASAT, ALAT, GGT, PAL, Bilirubin
Hepatomegaly | At Day 0 and Day 60
  liver damage evaluate by echography
C reactive protein | At Day 0, Day 30, Day 60
  Biological parameters to evaluate Systemic inflammation
sedimentation rate | At Day 0, Day 30, Day 60
  Biological parameters to evaluate Systemic inflammation
Immunoglobulin G level | At Day 0, Day 30, Day 60
  Biological parameters to evaluate Systemic inflammation
Haemoglobin level | At Day 0, Day 30, Day 60
  Biological parameters to evaluate inflammatory anaemia
Plasma concentration of methionine | From Day 0 to Day 75
  Variation of the concentration for each patient
Plasma concentration of homocysteine | From Day 0 to Day 75
  Variation of the concentration for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Alice HADCHOUEL, PhD, Principal Investigator — Hospital Necker Enfants Malades
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hadchouel A, Drummond D, Pontoizeau C, Aoust L, Hurtado Nedelec MM, El Benna J, Gachelin E, Perisson C, Vigier C, Schiff M, Lacaille F, Molina TJ, Berteloot L, Renolleau S, Ottolenghi C, Treluyer JM, de Blic J, Delacourt C. Methionine supplementation for multi-organ dysfunction in MetRS-related pulmonary alveolar proteinosis. Eur Respir J. 2022 Apr 21;59(4):2101554. doi: 10.1183/13993003.01554-2021. Print 2022 Apr. PMID 34503986